CLINICAL TRIAL: NCT03172442
Title: Dentoskeletal Effects of The Orthodontic Removable Traction Appliance in The Treatment of Skeletal Class III Malocclusion: A Randomized Controlled Trial
Brief Title: Treatment of Skeletal Class III Malocclusion Using Orthodontic Removable Traction Appliance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UDDS-Ortho-03-2017
Record Dates: First submitted 2017-05-23; First posted 2017-06-01 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Class III Malocclusion
Keywords: Class III treatment; orthodontic removable traction appliance; RCT
MeSH Terms: conditions — Malocclusion, Angle Class III

STUDY DESIGN:
Intervention Model Description: The patients will be randomly assigned to one of the two groups, case or control.
Masking Description: No masking could be applied
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- orthodontic removable traction appliance (Experimental): Patients in this group will be treated using the orthodontic removable traction appliance (vacuum plate with two hooks between lateral incisor and canine in each side). An rapid maxillary expander will be applied to disarticulate maxillary sutures to allow more efficient forward protraction of the maxilla.
  Class III elastic traction from upper first molar to the hook in both side. This appliance will be used full-time with Class III elastics (6- to 8-ounce) traction.
  Interventions: Device: Vacuum plate; Device: Rapid maxillary expander; Device: Class III elastics
- Control group (No Intervention): without intervention

INTERVENTIONS:
Device: Vacuum plate — Vacuum plate with two hooks between lateral incisor and canine in each side will be applied on the lower arch.
  Arms: orthodontic removable traction appliance
Device: Rapid maxillary expander — Rapid maxillary expander will be applied in the maxilla to disarticulate maxillary sutures to allow more efficient forward protraction of the maxilla.
  Arms: orthodontic removable traction appliance
Device: Class III elastics — Class III elastic traction from upper first molar to the hook in both side will be applied.
  Arms: orthodontic removable traction appliance

SUMMARY:
This experimental study aims to evaluate the efficiency of the orthodontic removable traction appliance in the treatment of skeletal class III malocclusion. The study sample will consist of 44 patients with skeletal class III malocclusion. The sample will be allocated randomly into two groups: experimental group and control group. The dentoskeletal changes will be assessed by using lateral cephalometric radiographs before treatment and after obtaining 3mm positive overjet.

DETAILED DESCRIPTION:
Treatment of class III malocclusion is a major challenge in orthodontic contemporary practice, Several appliance have suggested for the treatment of class III malocclusion, such as the facial mask and chin cup.

Despite of the efficiency of this extraoral appliance, its external appearance and its big size reduce patients' cooperation which decrease its clinical effects.

Another Class III treatment modality is the Orthodontic Removable Traction Appliance (ORTA). It is a removable appliance that can be used in conjunction with rapid palatal expansion or fixed appliances, It was developed in the 1980's by Dr. David Musich who developed this appliance in order to overcome issues of compliance that Dr. Musich experienced with use of the protraction facemask.

There is only one study that evaluated this appliance which is a retrospective study compared the treatment effects of the ORTA and protraction facemask in treatment of Class III malocclusions. However, this study has a lot of limitations which made it difficult to accurately evaluate the efficiency of this device.

The aim of this study is studying the dentoskeletal changes that result from treatment by this device, by comparing them to the changes in matched untreated group,by studying the cephalometric x-rays.

ELIGIBILITY:
Inclusion Criteria:

* Patients in early mixed dentation (8-10 years old).
* Skeletal class III caused by maxillary deficiency with or without mandibular prognathism judged clinically and confirmed radiographically(ANB≤1).
* Anterior crossbite on two teeth or more or an edge-to-edge bite.
* Normal inclination of the lower incisors with the mandibular plane.

Exclusion Criteria:

* Poor oral hygiene.
* Previous orthodontic treatment.
* Patients with syndromes, clefts, or craniofacial abnormalities.
* Severe skeletal class III primarily resulting from mandibular prognathism (ANB less than - 4)
* Patients with facial asymmetry.
* Patients with vertical growth pattern.

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2019-02-15 (Actual)

PRIMARY OUTCOMES:
The change of the ANB angle | Assessment will be done before treatment (T0) and after obtaining 3-mm positive overjet which will be approximately obtained after 6 months (T1).
  The change of the ANB angle before and after using the Orthodontic Removable Traction Appliance compared with this of the control group will be evaluated using lateral cephalometric radiographs.

SECONDARY OUTCOMES:
The change of the SNA angle | Assessment will be done before treatment (T0) and after obtaining 3-mm positive overjet which will be approximately obtained after 6 months (T1).
  The change of the SNA angle before and after using the Orthodontic Removable Traction Appliance compared with this of the control group will be evaluated using lateral cephalometric radiographs.
The change of the SNB angle | Assessment will be done before treatment (T0) and after obtaining 3-mm positive overjet which will be approximately obtained after 6 months (T1).
  The change of the SNB angle before and after using the Orthodontic Removable Traction Appliance compared with this of the control group will be evaluated using lateral cephalometric radiographs.
Levels of pain | A questionnaire will be given to the patients four times during treatment; after 1day, after 1 week, after 1 month and after 3 months of the application of the appliance.
  The level of Pain caused by using the Orthodontic Removable Traction Appliance will be assessed using a questionnaire with a Visual Analog Scale (VAS).
Levels of discomfort | A questionnaire will be given to the patients four times during treatment; after 1day, after 1 week, after 1 month and after 3 months of the application of the appliance.
  The level of discomfort caused by using the Orthodontic Removable Traction Appliance will be assessed using a questionnaire with a Visual Analog Scale (VAS).
Levels of acceptance | A questionnaire will be given to the patients four times during treatment; after 1day, after 1 week, after 1 month and after 3 months of the application of the appliance.
  The level of acceptance of using the Orthodontic Removable Traction Appliance will be assessed using a questionnaire with a Visual Analog Scale (VAS).

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad S Burhan, PhD., Study Chair — Department of Orthodontics, Faculty of Dentistry, Damascus University, Damascus, Syria
Locations (1):
- Damascus University, Damascus, Syria

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be available to the researchers in the department of Orthodontics, Damascus University

REFERENCES:
- [Result] Cha KS. Skeletal changes of maxillary protraction in patients exhibiting skeletal class III malocclusion: a comparison of three skeletal maturation groups. Angle Orthod. 2003 Feb;73(1):26-35. doi: 10.1043/0003-3219(2003)0732.0.CO;2. PMID 12607852
- [Result] Mandall N, DiBiase A, Littlewood S, Nute S, Stivaros N, McDowall R, Shargill I, Worthington H, Cousley R, Dyer F, Mattick R, Doherty B. Is early Class III protraction facemask treatment effective? A multicentre, randomized, controlled trial: 15-month follow-up. J Orthod. 2010 Sep;37(3):149-61. doi: 10.1179/14653121043056. PMID 20805344
- [Result] Gautam P, Valiathan A, Adhikari R. Skeletal response to maxillary protraction with and without maxillary expansion: a finite element study. Am J Orthod Dentofacial Orthop. 2009 Jun;135(6):723-8. doi: 10.1016/j.ajodo.2007.06.016. PMID 19524831
- [Result] Turley PK. Orthopedic correction of Class III malocclusion with palatal expansion and custom protraction headgear. J Clin Orthod. 1988 May;22(5):314-25. No abstract available. PMID 3075214
- [Result] Suda N, Ishii-Suzuki M, Hirose K, Hiyama S, Suzuki S, Kuroda T. Effective treatment plan for maxillary protraction: is the bone age useful to determine the treatment plan? Am J Orthod Dentofacial Orthop. 2000 Jul;118(1):55-62. doi: 10.1067/mod.2000.104491. PMID 10893473